CLINICAL TRIAL: NCT02460835
Title: A Pilot Study of Individualized Adaptive Radiation Therapy for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.039; HUM00098022 (Other: University of Michigan)
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adaptive Radiation Therapy (Experimental)
  Interventions: Radiation: Adaptive Radiation Therapy

INTERVENTIONS:
Radiation: Adaptive Radiation Therapy

SUMMARY:
This is a pilot single arm study with the primary endpoints of feasibility and preliminary estimates of safety and efficacy. This protocol builds on over 25 years of experience with high dose liver RT (Radiation Therapy), and in particular adaptive RT aimed at adjusting the global radiation dose based on a patient's measured sensitivity to treatment. This current protocol uses functional imaging and specialized radiation planning techniques to spare highly functional portions of the liver to preserve function. The investigators feel this will further improve the safety and efficacy of RT for all patients by customizing treatments to each. If this approach is promising, the investigators will proceed to a phase II randomized study of standard versus spatially and dosimetrically adapted RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have hepatocellular carcinoma.
* Patients must not have extrahepatic cancer.
* Patients must not be eligible for a curative liver resection or have refused resection
* Patients must have recovered from the acute effects of prior liver-directed therapy and 4 weeks must have passed since the last procedure and protocol therapy.
* Patients must have a Zubrod performance status of less than or equal to 2 (Zubrod performance status is a measure that attempts to quantify a cancer patients' general well-being. Scores run from 0 to 5 where 0 denotes normal activity and 5 denotes death).
* Patients must be 18 years of age or older.
* Patients must have adequate organ function.
* Patients must understand and be willing to sign an IRB (Institutional Review Board) approved informed consent form.

Exclusion Criteria:

* Patients with known allergies to intravenous iodinated contrast agents.
* Patients with a contraindication to contrast-enhanced MRI are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Lawrence, M.D., Ph.D., Principal Investigator — Rogel Cancer Center
Locations (1):
- Rogel Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Adaptive Radiation Therapy: Adaptive Radiation Therapy
Period: Overall Study
Arm/Group | Adaptive Radiation Therapy
Started | 77
Completed | 56
Not Completed | 21
Not completed — Disease progression prior to treatment | 3
Not completed — Unable to complete planning scans | 2
Not completed — Decrease in performance status | 1
Not completed — Withdrawal by Subject | 3
Not completed — Underwent fractionated RT | 10
Not completed — Unable to complete follow-up lab draws | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 35
Age, Continuous [Mean (Full Range); unit: years] | 63 [48 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 68
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients for Whom the Intended Treatment Was Feasible
Description: The primary aim of the trial is feasibility which is defined as the ability to successfully deliver the full treatment including all adaptations and in particular the perfusion-based planning and replanning.
Time Frame: At end of treatment; up to ~3 months
Population: 77 subjects enrolled, 70 subjects treated
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 77
Participants | 70

2. Primary Outcome: Percentage of Patients With Change in Child Pugh Score >= 2
Description: Rate of liver decompensation reported as the percentage of patients with a change in Child Pugh score of greater than or equal to 2 within 6 months of SBRT.
Time Frame: Baseline to approximately 6 months after initiation of SBRT
Population: 77 subjects enrolled, 70 subjects treated, 56 eligible for analysis (14 were excluded: 10- fractionated RT, 2- unable to complete follow up, 2- withdrew)
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 56
Participants | 12

3. Primary Outcome: Median Time to Local Progression
Description: The primary efficacy endpoint is local control, measured as the duration of time from start of treatment to time of progression of the treated (target) lesion(s). Patients with no evidence of local progression at the time of data analysis will be censored at the last date on which they were evaluated for local progression. Local progression will be summarized with Kaplan-Meier curves and reported with 95% confidence intervals.
Time Frame: 24 months
Population: 77 subjects enrolled, 70 subjects treated, 9 eligible for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 9
Months | 17.4 [4.93 to 25.27]

4. Secondary Outcome: Median Time to Progression
Description: Defined as the duration of time from start of treatment to time of progression.
Time Frame: 24 months
Population: 77 subjects enrolled, 70 subjects treated, 31 eligible for analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 31
months | 5.23 [4.57 to 9.03]

5. Secondary Outcome: Change in ALBI Scores
Description: Liver decompensation assessed by change in ALBI score > 0.5 from baseline.
Time Frame: Approximately 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 56
Participants | 15

6. Secondary Outcome: Incidence of Grade 3 Gastrointestinal (GI) Bleeding Toxicities
Description: Grade 3 GI bleeding assessed via the NCI CTCAE version 4.0.
Time Frame: Approximately 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 56
Participants | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the duration of time from start of treatment to death.
Time Frame: 24 months
Population: 77 subjects enrolled, 70 subjects treated, 54 eligible for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adaptive Radiation Therapy
Number analyzed (Participants) | 54
Months | 16.8 [10.67 to 28.47]

8. Other Pre Specified Outcome: Incidence of Radiation Induced Liver Disease (RILD)
Description: RILD is a rare but serious side effect that will be summarized if it occurs.
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 2 years after last dose of study treatment. Data was collected over 6 years.
Arm/Group | Adaptive Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 19/77
Serious Adverse Events (participants affected / at risk) | 6/77
Other Adverse Events (participants affected / at risk) | 67/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive Radiation Therapy (N=77)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Catheter Related Infection (Infections and infestations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive Radiation Therapy (N=77)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 7 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 6 (6)
Chills (General disorders) | 1 (1)
Edema Limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 31 (34)
Multi-organ Failure (General disorders) | 1 (1)
Hepatic Pain (Hepatobiliary disorders) | 5 (5)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood Bilirubin increased (Investigations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
dizziness (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT02460835/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT02460835/ICF_001.pdf